CLINICAL TRIAL: NCT03112850
Title: Investigating the Impact of Hearing Aid Use and Auditory Training on Cognition, Mood and Social Interaction in Older Adults With Hearing Loss
Brief Title: Cognition Effects of Hearing Aids and Auditory Training in Older Age
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swinburne University of Technology (Other)
Responsible Party: Principal Investigator, Denny Meyer, Professor, Swinburne University of Technology
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SHR Project 2016/159
Record Dates: First submitted 2017-04-01; First posted 2017-04-13 (Actual); Last update posted 2018-09-07 (Actual); Status verified 2018-09

CONDITIONS: Hearing Loss, Sensorineural
Keywords: Crossover design; Randomized controlled trial; Aural rehabilitation intervention
MeSH Terms: conditions — Hearing Loss, Sensorineural | interventions — Hearing Aids

STUDY DESIGN:
Intervention Model Description: This is a randomised crossover trial with participants randomized into two equal groups to carry out separate crossover experiments. All participants will undergo an individualised auditory training for a period of 6 months, and will be randomly allocated to one of the following groups.
  1. Participants who will be fitted with hearing aids for the first 3 months of auditory training program - Group A
  2. Participants who will be fitted with hearing aids for the last 3 months of auditory training program - Group B Groups will be matched in terms of the degree of hearing loss with one member from each matched pair randomly assigned to Group A and the other member of each matched pair assigned to Group B. A random sequence of binary digits will be used for this purpose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): Participants who will be fitted with hearing aids for the first 3 months of 6 months auditory training program
  Interventions: Device: Hearing aid; Behavioral: Auditory Training
- Group B (Active Comparator): Participants who will be fitted with hearing aids for the second 3 months of 6 months auditory training program
  Interventions: Device: Hearing aid; Behavioral: Auditory Training

INTERVENTIONS:
Device: Hearing aid — LOF hearing aid
Behavioral: Auditory Training

SUMMARY:
Sensorineural type of hearing loss is the most common sensory deficit among older adults. Some of the psychosocial consequences of this condition include difficulty in understanding speech, depression and social isolation. Studies have shown that older adults with hearing loss show some age-related cognitive decline. There is no clinically proven method to predict the onset of this condition, as its occurrence is slow and progressive, affecting both ears equally. Although hearing aid use and auditory training have been proven as successful interventions to alleviate sensorineural hearing loss, no research has been designed to look at the effect of both hearing aid use coupled with auditory training on cognitive performance in older adults. This study will investigate whether wearing hearing aids will improve the impact of auditory training on cognition, mood and social interaction for older adults with sensorineural hearing loss.

This is a crossover trial targeting older adults between 50 and 90 years with either mild or moderate symmetric sensorineural hearing loss. Consented, willing participants will undergo a six month intensive auditory training program (active control), as a rigorous means of examining the impact hearing aid use has on a person's cognition, mood and social interaction. Participants will be assigned in random order to receive hearing aid (intervention) for either the first three or last three months of the six month auditory training program. Each participant will be tested at baseline, three and six months on a battery of computer based cognitive assessments, together with mood, and social engagement measures. Effectiveness of hearing aids and auditory training will be evaluated using an online speech perception test (SPT) and the Abbreviated Profile of Hearing Aid Benefit (APHAB) Inventory.

This study will investigate whether using a hearing aid coupled with auditory training can improve a person's cognition and learning abilities, relationships with family and friends, and quality of life. Results from the study will inform strategies for aural rehabilitation, hearing aid delivery and future hearing loss intervention trials.

DETAILED DESCRIPTION:
Background:

Sensorineural hearing loss is the most common sensory deficit among older adults. There is no clinically proven method to predict the onset of this condition, as its occurrence is generally slow and progressive, affecting both ears equally. Recent studies have documented that hearing loss in older adults is independently associated with reduced cognitive functioning, mood and social interaction, and that hearing aid use and auditory training could improve cognitive abilities, social, emotional, psychological, and physical well-being of people. Despite the high prevalence of hearing loss in older adults, and the consequences for health outcomes, people are generally slow to acquire hearing aids, and almost two-thirds of older adults with hearing impairment do not use hearing aids. The popularity of auditory training has also declined in recent years and the focus of research has been shifted to only improving wearable amplification such as hearing aids. No research has been designed to specifically look at the effect of both hearing aid use coupled with auditory training on cognitive performance in older adults.

Study aim:

The aim of the current study is to investigate the impact of hearing aid use coupled with auditory training on mood, social relationships and cognitive functioning in a crossover intervention trial.

Study hypothesis:

The rationale for this study objective is based on the following hypotheses:

H1: In older adults with sensorineural hearing loss, hearing aids in combination with auditory training will be more effective for improving cognition than auditory training on its own.

H2: In older adults with sensorineural hearing loss, hearing aids in combination with auditory training will be more effective for improving mood and social interaction than auditory training on its own.

Crossover design:

This is a randomised crossover trial with a total of 40 participants randomized into two equal groups (20 each) to carry out separate crossover experiments. All participants will undergo individualised auditory training for a period of 6 months, and will be randomly allocated to one of the following groups.

1. Participants who will be fitted with hearing aids only for the first 3 months of the auditory training program - Group A
2. Participants who will be fitted with hearing aids only for the last 3 months of the auditory training program - Group B Participants will be tested at baseline, and at three and six months in terms of cognition, mood and social engagement. The primary outcome measure will be changes in cognitive performance as measured by the Swinburne University Computerized Assessment Battery (SUCCAB). Secondary outcome measures will include changes in mood and social engagement scores.

Setting of the study This study is set in Victoria, Australia. It will be conducted in independent living aged care facilities across Melbourne. These residents live in their own unit or similar accommodation, and are generally capable of caring for themselves in all aspects of daily living. In addition, elderly participants from the Swinburne University of Technology's Centre for Human Psychopharmacology (CHP) database who live independently will be recruited to take part in the study.

Recruitment:

Independent living aged care facilities will be contacted by telephone to explain the study. If an aged care facility shows interest in the study, researchers will visit the facility to provide the facility manager with more detailed written and oral information. If the facility manager consents for their facility to participate in the study, the study will be advertised at the facility and flyers will be distributed to all the residents inviting them to an information session. Participants from the Swinburne University of Technology's CHP database will be contacted by telephone and email to explain the study and participants who express interest will be invited to attend an information session. At the information session, researchers will explain the purpose and significance of the study. At the same time, a pre-selection screening will be conducted to identify participants who are cognitively healthy, likely to benefit from hearing rehabilitation, and who will be able to participate in the cognition battery testing (reasonable sight and not colour blind). Selected participants will be sent a Participant Information and Consent Form package that includes detailed information on the study procedure, a consent form and a return pre-paid envelope. Once written consent is received, participants will be invited to complete baseline measures and to confirm their eligibility before enrolment into the study.

Participants:

The baseline cohort will consist of forty (40) older adults with either a mild or moderate symmetric sensorineural hearing loss. All participants will be first time hearing aid users, having never worn hearing aids previously. Participants will be screened for adequate cognitive functioning using the Mini-mental state examination (MMSE). Participants must have a global cognitive impairment as determined by a score greater than 24 on the (MMSE).

Sample size:

Power analyses were conducted to determine the sample size required. Previous research and the results of the power analysis suggest that a total sample size of 36 is sufficient to detect a moderate size effect (f=0.25), with power of 80% and a significance level of 5%. Therefore, a total sample size of 40 participants will be recruited to provide a definitive test of the hypotheses, while allowing for 10% attrition.

Data collection methods:

The assessments selected for this study are categorized as:

1. Hearing Assessments

   * Otoscopy and tympanometry: Following otoscopy, all participants will undergo tympanometry and acoustic reflex testing to assess the status of the middle ear.
   * Pure tone audiometry in each ear: To understand the degree of hearing impairment, hearing ability will be measured at threshold frequencies 0.5, 1, 2, 3, 4, 6 kHz in both ears. An online Speech Perception Test will be used in addition to the standard audiograms for the purpose of measuring hearing loss and hearing aid fitting.
2. Paper-based Questionnaire

Participants will complete a paper-based questionnaire which will be structured in the following sections:

* Demographics: Information on a variety of demographic variables will be collected in order to describe the characteristics of the study participants
* The Geriatric Depression Scale (GDS): To assess mood, the short version of the GDS will be used to detect the depressive symptoms in the elderly.
* Social Engagement Measure: The Berkman-Syme Social Network Index will be used to measure participants' social engagement and connections with families, friends, etc.
* The Mini-Mental State Examination (MMSE) Questionnaire: The MMSE will be used as a screening criterion to assess cognition.

  3. Cognitive Assessments
* The Swinburne University Computerized Assessment Battery (SUCCAB) will be used as a primary measure to assess cognitive performance. Reliability and validity testing of this battery has demonstrated that the SUCCAB is sensitive to ageing, and has been shown to be particularly effective for measuring short-term changes in cognition for the elderly. The SUCCAB correlates strongly with memory subsets in the Wechsler Adult Intelligence Scales.

All participants who will be enrolled into the study will complete these assessments again at 3 months and at 6 months.

Interventions:

Fitting of hearing aids for Group A and Group B participants:

Participants will be fitted with two Blamey Saunders hearing aids known as the LOF for a period of 3 months. The hearing aids will be fitted according to the manufacturer's protocol, and explanation of the hearing aid usage, insertion of the aids and batteries along with a step-by-step guide on how to use the hearing aid will be given. A data logging function in the hearing aids will be used to assess hours of hearing aid use.

After 3 months (with wearing their hearing aids)

In addition, the Abbreviated Profile of Hearing Aid Benefit (APHAB), a self-assessment inventory, will be carried out with the assistance of the researcher to assess hearing aid benefit. Four scales of the APHAB will be assessed namely:

* Ease of communication (EC)
* Effects of background noise (BN)
* Effects of reverberation (RV), such as listening to sounds across a large room Aversiveness (AV), which will look at uncomfortable loudness of background sounds such as traffic and alarm bells.

Auditory training:

All participants enrolled into the study will undergo weekly auditory training for a period of 6 months. Over the 6 month period, each participant will undergo a two 12-week individualised speech tracking program, called the Continuous Discourse Speech Tracking, with and without hearing aids. Each test session will last for approximately 15 minutes. The procedure will be timed and scored in number of words per minute (wpm) transmitted. Tracking rate will be calculated as the number of words correctly repeated divided by the time elapsed.

Working Alliance Inventory:

At the end of the 6 month period after all examinations have been completed, Group A and B participants will complete a working alliance inventory, in order to evaluate the following: the quality of participant-researcher relationship, the collaborative nature of agreeing on tasks and goals of both auditory training and hearing aid compliance, and the outcome measures from auditory training provided to participants. Some randomized controlled trials have demonstrated that this evaluation is crucial for engaging, retaining and improving positive outcomes for study participants, and is vital for relationship-building.

Planned analysis

* Baseline comparison of the two groups in terms of demographics, cognition, mood, social engagement, hearing loss and hearing satisfaction using appropriate chi-square test, t-test and non-parametric Mann-Whitney tests.
* Comparison of the two groups in terms of changes in cognition, mood, social engagement from baseline to 3 months and 6 months, using a crossover analysis and multi-level models, allowing for any carry-over effect.
* The analysis of speech perception test results with and without hearing aids as a measure of the effectiveness of hearing aids and auditory training with and without hearing aids using multi-level models and again allowing for carry-over effects.
* The speech tracking rates from the two 12-week programs of speech tracking will be analysed for each participant using a learning model. This analysis will yield learning and forgetting rates with and without hearing aids. These learning and forgetting rates are valid measures of cognitive processes that are likely to be affected by the use of hearing and hearing aids. This data will also be analysed using multi-level models and again allowing for carry-over effects.

Contingency Plan: For participants who decide to discontinue auditory training because hearing aids have been beneficial, or decide to drop out entirely in the course of the auditory training program, they will be retained in the study as a third group, with a suitable modification to the analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged between 50 and 90 years
2. Have good working knowledge of English
3. Mild or moderate symmetric sensorineural hearing loss with a pure-tone average (PTA) of thresholds at 0.5 - 6 kHz in both ears
4. Willing to wear hearing aids for three (3) months
5. Willing to undergo weekly auditory training for a period of six (6) months.
6. Submit written consent to participant in study

Exclusion Criteria:

1. Any significant visual impairment that would prevent them from reading or performing computer based tasks.
2. Suspected cognitive impairment (defined as a score less or equal to 24 on the MMSE)
3. Severe or profound hearing loss

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change over six months in SUCCAB performance (accuracy/reaction time) measures | Change from baseline to six months
  The SUCCAB contains a battery of eight cognitive domains namely Simple and Choice Reaction Times, Immediate and Delayed Recognition, Congruent and Incongruent Stroop colour-words, Spatial Working Memory and Contextual Memory.

SECONDARY OUTCOMES:
Change in the Geriatric Depression Scale (GDS) aggregated into a single score | Change from baseline to six months
  The GDS is a self-rating screening scale for depression in the elderly population. To assess mood, the short version of the GDS will be used to detect the depressive symptoms in the elderly
The Berkman-Syme Social Network Index aggregated into a single score | Change from baseline to six months
  The Berkman-Syme Social Network Index will be used to assess participant's social engagement and connections with families and friends

CONTACTS AND LOCATIONS:
Overall Officials: Denny Meyer, PhD, Principal Investigator — Swinburne University of Technology
Locations (1):
- Swinburne University of Technology, Melbourne, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided
There is no plan

REFERENCES:
- [Background] Gates GA, Mills JH. Presbycusis. Lancet. 2005 Sep 24-30;366(9491):1111-20. doi: 10.1016/S0140-6736(05)67423-5. PMID 16182900
- [Background] Murphy CF, Fillippini R, Palma D, Zalcman TE, Lima JP, Schochat E. Auditory training and cognitive functioning in adult with traumatic brain injury. Clinics (Sao Paulo). 2011;66(4):713-5. doi: 10.1590/s1807-59322011000400030. No abstract available. PMID 21655770
- [Background] Amieva H, Ouvrard C, Giulioli C, Meillon C, Rullier L, Dartigues JF. Self-Reported Hearing Loss, Hearing Aids, and Cognitive Decline in Elderly Adults: A 25-Year Study. J Am Geriatr Soc. 2015 Oct;63(10):2099-104. doi: 10.1111/jgs.13649. PMID 26480972
- [Background] Lin FR, Yaffe K, Xia J, Xue QL, Harris TB, Purchase-Helzner E, Satterfield S, Ayonayon HN, Ferrucci L, Simonsick EM; Health ABC Study Group. Hearing loss and cognitive decline in older adults. JAMA Intern Med. 2013 Feb 25;173(4):293-9. doi: 10.1001/jamainternmed.2013.1868. PMID 23337978
- [Background] Davis A, Smith P, Ferguson M, Stephens D, Gianopoulos I. Acceptability, benefit and costs of early screening for hearing disability: a study of potential screening tests and models. Health Technol Assess. 2007 Oct;11(42):1-294. doi: 10.3310/hta11420. PMID 17927921
- [Background] Fischer ME, Cruickshanks KJ, Wiley TL, Klein BE, Klein R, Tweed TS. Determinants of hearing aid acquisition in older adults. Am J Public Health. 2011 Aug;101(8):1449-55. doi: 10.2105/AJPH.2010.300078. Epub 2011 Jun 16. PMID 21680930
- [Background] Folstein MF, Folstein SE, McHugh PR. "Mini-mental state". A practical method for grading the cognitive state of patients for the clinician. J Psychiatr Res. 1975 Nov;12(3):189-98. doi: 10.1016/0022-3956(75)90026-6. No abstract available. PMID 1202204
- [Background] Acar B, Yurekli MF, Babademez MA, Karabulut H, Karasen RM. Effects of hearing aids on cognitive functions and depressive signs in elderly people. Arch Gerontol Geriatr. 2011 May-Jun;52(3):250-2. doi: 10.1016/j.archger.2010.04.013. Epub 2010 May 15. PMID 20472312
- [Background] Blamey PJ, Blamey JK, Saunders E. Effectiveness of a teleaudiology approach to hearing aid fitting. J Telemed Telecare. 2015 Dec;21(8):474-8. doi: 10.1177/1357633X15611568. PMID 26556060
- [Background] Burke WJ, Roccaforte WH, Wengel SP. The short form of the Geriatric Depression Scale: a comparison with the 30-item form. J Geriatr Psychiatry Neurol. 1991 Jul-Sep;4(3):173-8. doi: 10.1177/089198879100400310. PMID 1953971
- [Background] Berkman LF, Syme SL. Social networks, host resistance, and mortality: a nine-year follow-up study of Alameda County residents. Am J Epidemiol. 1979 Feb;109(2):186-204. doi: 10.1093/oxfordjournals.aje.a112674. PMID 425958
- [Background] Hardman RJ, Kennedy G, Macpherson H, Scholey AB, Pipingas A. A randomised controlled trial investigating the effects of Mediterranean diet and aerobic exercise on cognition in cognitively healthy older people living independently within aged care facilities: the Lifestyle Intervention in Independent Living Aged Care (LIILAC) study protocol [ACTRN12614001133628]. Nutr J. 2015 May 24;14:53. doi: 10.1186/s12937-015-0042-z. PMID 26003546
- [Background] Cox RM, Alexander GC. The abbreviated profile of hearing aid benefit. Ear Hear. 1995 Apr;16(2):176-86. doi: 10.1097/00003446-199504000-00005. PMID 7789669
- [Background] De Filippo CL, Scott BL. A method for training and evaluating the reception of ongoing speech. J Acoust Soc Am. 1978 Apr;63(4):1186-92. doi: 10.1121/1.381827. PMID 649877
- [Background] Cunningham PB, Henggeler SW. Engaging multiproblem families in treatment: lessons learned throughout the development of multisystemic therapy. Fam Process. 1999 Fall;38(3):265-81. doi: 10.1111/j.1545-5300.1999.00265.x. PMID 10526764
- [Background] Liddle HA, Dakof GA, Parker K, Diamond GS, Barrett K, Tejeda M. Multidimensional family therapy for adolescent drug abuse: results of a randomized clinical trial. Am J Drug Alcohol Abuse. 2001 Nov;27(4):651-88. doi: 10.1081/ada-100107661. PMID 11727882
- [Derived] Nkyekyer J, Meyer D, Blamey PJ, Pipingas A, Bhar S. Investigating the Impact of Hearing Aid Use and Auditory Training on Cognition, Depressive Symptoms, and Social Interaction in Adults With Hearing Loss: Protocol for a Crossover Trial. JMIR Res Protoc. 2018 Mar 23;7(3):e85. doi: 10.2196/resprot.8936. PMID 29572201